CLINICAL TRIAL: NCT03227471
Title: A Phase 1/2 Study of VX-445 in Healthy Subjects and Subjects With Cystic Fibrosis
Brief Title: A Study of VX-445 in Healthy Subjects and Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX16-445-001; 2017-000797-11 (EudraCT Number)
Record Dates: First submitted 2017-07-18; First posted 2017-07-24 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor; tezacaftor, ivacaftor drug combination; elexacaftor; tezacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Part A: Pooled Placebo (Except Cohort A7) (Placebo Comparator): Participants without CF who received single dose of placebo matched to VX-445 in Cohort A1 to A5.
  Interventions: Drug: Matched Placebo
- Part A: VX-445 (Except Cohort A7) (Experimental): Participants without CF who received single ascending dose of VX-445 tablet starting from 20 milligrams (mg) to 360 mg in Cohort A1 to A5.
  Interventions: Drug: VX-445
- Part A: VX-445 (Cohort A7) (Experimental): Participants without CF who received single dose of VX-445 100 mg tablet on Day 1 in fasted state and on Day 7 in fed state, followed by VX-445 20 mg intravenous (IV) injection on Day 13 in fed state in Cohort A7.
  Interventions: Drug: VX-445
- Part B: Pooled Placebo (Cohort B1 to B4) (Placebo Comparator): Participants without CF who received multiple doses of placebo matched to VX-445 once daily (qd) for 10 days in Cohort B1 to B4.
  Interventions: Drug: Matched Placebo
- Part B: VX-445 (Cohort B1 to B4) (Experimental): Participants without CF who received VX-445 tablet qd for 10 days in Cohort B1 (60 mg), B2 (120 mg), B3 (240 mg) and B4 (340 mg).
  Interventions: Drug: VX-445
- Part C: Pooled Placebo (Cohort C1 to C3) (Placebo Comparator): Participants without CF who received placebo matched to VX-445/TEZ/IVA triple combination (TC) qd in the morning and placebo matched to IVA in the evening for 14 days.
  Interventions: Drug: Matched Placebo
- Part C: VX-445/TEZ/IVA TC (Cohort C1 to C3) (Experimental): Participants without CF who received VX-445 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in Cohort C1; VX-445 280 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in Cohort C2 and VX-445 100 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in Cohort C3 for 14 days.
  Interventions: Drug: IVA; Drug: TEZ/IVA; Drug: VX-445
- Part D: Placebo (Placebo Comparator): Participants with CF, F/MF genotype who received placebo matched to VX-445/TEZ/IVA TC qd in the morning and placebo matched to IVA qd in the evening for 4 weeks in the TC treatment period.
  Interventions: Drug: Matched Placebo
- Part D: VX-445/TEZ/IVA TC - Low Dose (Experimental): Participants with CF, F/MF genotype who received VX-445 50 mg qd/TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the TC treatment period.
  Interventions: Drug: IVA; Drug: TEZ/IVA; Drug: VX-445
- Part D: VX-445/TEZ/IVA TC - Medium Dose (Experimental): Participants with CF, F/MF genotype who received VX-445 100 mg qd/TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the TC treatment period.
  Interventions: Drug: IVA; Drug: TEZ/IVA; Drug: VX-445
- Part D: VX-445/TEZ/IVA TC - High Dose (Experimental): Participants with CF, F/MF genotype who received VX-445 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the TC treatment period.
  Interventions: Drug: IVA; Drug: TEZ/IVA; Drug: VX-445
- Part E: TEZ/IVA (Active Comparator): Following run-in period of 4 weeks with TEZ/IVA, participants with CF, F/F genotype who received TEZ 100 mg qd/IVA 150 mg q12h and placebo matched to VX-445 for 4 weeks in the TC treatment period.
  Interventions: Drug: TEZ/IVA
- Part E: VX-445/TEZ/IVA TC (Experimental): Following run-in period of 4 weeks with TEZ/IVA, participants with CF, F/F genotype who received VX-445 200 mg qd/TEZ 100 mg qd /IVA 150 mg q12h for 4 weeks in the TC treatment period.
  Interventions: Drug: IVA; Drug: TEZ/IVA; Drug: VX-445
- Part F: Placebo (Placebo Comparator): Participants with CF, F/MF genotype who received placebo matched to VX-445/TEZ/VX-561 for 4 weeks in the TC treatment period.
  Interventions: Drug: Matched Placebo
- Part F: VX-445/TEZ/VX-561 TC (Experimental): Participants with CF, F/MF genotype who received VX-445 200 mg qd/TEZ 100 mg qd/VX-561 150 mg qd for 4 weeks in the TC treatment period.
  Interventions: Drug: VX-445; Drug: TEZ; Drug: VX-561

INTERVENTIONS:
Drug: IVA — IVA tablet for oral administration
  Other Names: VX-770; ivacaftor
  Arms: Part C: VX-445/TEZ/IVA TC (Cohort C1 to C3); Part D: VX-445/TEZ/IVA TC - High Dose; Part D: VX-445/TEZ/IVA TC - Low Dose; Part D: VX-445/TEZ/IVA TC - Medium Dose; Part E: VX-445/TEZ/IVA TC
Drug: TEZ/IVA — TEZ/IVA fixed-dose combination for oral administration.
  Other Names: VX-661/VX-770; tezacaftor/ivacaftor
  Arms: Part C: VX-445/TEZ/IVA TC (Cohort C1 to C3); Part D: VX-445/TEZ/IVA TC - High Dose; Part D: VX-445/TEZ/IVA TC - Low Dose; Part D: VX-445/TEZ/IVA TC - Medium Dose; Part E: TEZ/IVA; Part E: VX-445/TEZ/IVA TC
Drug: VX-445 — VX-445 tablet for oral administration.
  Other Names: ELX; elexacaftor
  Arms: Part A: VX-445 (Cohort A7); Part A: VX-445 (Except Cohort A7); Part B: VX-445 (Cohort B1 to B4); Part C: VX-445/TEZ/IVA TC (Cohort C1 to C3); Part D: VX-445/TEZ/IVA TC - High Dose; Part D: VX-445/TEZ/IVA TC - Low Dose; Part D: VX-445/TEZ/IVA TC - Medium Dose; Part E: VX-445/TEZ/IVA TC; Part F: VX-445/TEZ/VX-561 TC
Drug: Matched Placebo — Matched placebo.
  Arms: Part A: Pooled Placebo (Except Cohort A7); Part B: Pooled Placebo (Cohort B1 to B4); Part C: Pooled Placebo (Cohort C1 to C3); Part D: Placebo; Part F: Placebo
Drug: TEZ — Tablet for oral administration.
  Other Names: VX-661; tezacaftor
  Arms: Part F: VX-445/TEZ/VX-561 TC
Drug: VX-561 — Tablet for oral administration.
  Other Names: CTP-656
  Arms: Part F: VX-445/TEZ/VX-561 TC
Drug: VX-445 — VX-445 IV injection
  Other Names: ELX; elexacaftor
  Arms: Part A: VX-445 (Cohort A7)

SUMMARY:
This is a first-in-human and proof-of-concept study of VX-445. The study includes 6 parts. Parts A, B, and C were conducted in healthy subjects. Parts D, E, and F were conducted in subjects with Cystic Fibrosis (CF) who are homozygous for the F508del mutation of the CF transmembrane conductance regulator (CFTR) gene (F/F genotype), or who are heterozygous for the F508del mutation and a minimal function (MF) CFTR mutation not likely to respond to TEZ, IVA, or TEZ/IVA (F/MF genotypes).

ELIGIBILITY:
Key Inclusion Criteria:

Parts A, B, and C:

* Female subjects must be of non-childbearing potential.
* Between the ages of 18 and 55 years, inclusive.
* Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive, and a total body weight >50 kg

Parts D, E, and F:

* Body weight ≥35 kg.
* Subjects must have an eligible CFTR genotype:

  * Parts D and F: Heterozygous for F508del and an MF mutation (F/MF)
  * Part E: Homozygous for F508del (F/F)
* FEV1 value ≥40% and ≤90% of predicted mean for age, sex, and height.

Key Exclusion Criteria:

Parts A, B, and C:

* Any condition possibly affecting drug absorption.
* History of febrile illness within 14 days before the first study drug dose.
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency.

Parts D, E, and F:

* History of clinically significant cirrhosis with or without portal hypertension.
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Lung infection with organisms associated with a more rapid decline in pulmonary status.
* History of solid organ or hematological transplantation.

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (26):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Valley Children's Healthcare, Madera, California
  - (Kaiser Permanente) Oakland Medical Center, Oakland, California
  - National Jewish Health, Denver, Colorado
  - Central Florida Pulmonary Group, Orlando, Florida
  - Tampa General Hospital Cardiac and Lung Transplant Clinic, Tampa, Florida
  - Children's Specialty Services at North Druid Hills, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Covance Clinical Research Unit Inc., Evansville Clinic [Parts A, B, C only], Evansville, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane Medical Center, New Orleans, Louisiana
  - Harper University Hospital, Detroit, Michigan
  - Children's Respiratory and Critical Care Specialists, P.A., Children's Hospitals and Clinics of Minn, Minneapolis, Minnesota
  - Morristown Medical Center, Morristown, New Jersey
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - UC Health Office of Clinical Research, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center/Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Austin Children's Chest Associates, Austin, Texas
  - The University of Vermont, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - West Virginia University Hospitals, Morgantown, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - Monash Medical Center, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Children's Hospital Melbourne, Parkville, Victoria
  - Mater Adult Hospital, Brisbane
  - Royal Prince Alfred Hospital, Sydney
  - Westmead Hospital, Sydney
- Belgium (2):
  - Antwerp University Hospital, Edegem
  - Universitair Ziekenhuis Gent, Ghent
- Netherlands (4):
  - Academic Medical Centre, Amsterdam
  - Radboud UMC, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis van den Haag, The Hague

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- [Derived] Keating D, Marigowda G, Burr L, Daines C, Mall MA, McKone EF, Ramsey BW, Rowe SM, Sass LA, Tullis E, McKee CM, Moskowitz SM, Robertson S, Savage J, Simard C, Van Goor F, Waltz D, Xuan F, Young T, Taylor-Cousar JL; VX16-445-001 Study Group. VX-445-Tezacaftor-Ivacaftor in Patients with Cystic Fibrosis and One or Two Phe508del Alleles. N Engl J Med. 2018 Oct 25;379(17):1612-1620. doi: 10.1056/NEJMoa1807120. Epub 2018 Oct 18. PMID 30334692

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included 6 parts: Parts A, B, and C were conducted in healthy adult participants; Part D, E, and F were conducted in adult cystic fibrosis (CF) participants.
Groups:
- Part B: VX-445 (Cohort B1 to B4): Participants without CF who received VX-445 tablet once daily for 10 days in Cohort B1 (60 mg), B2 (120 mg), B3 (240 mg) and B4 (340 mg).
- Part C: Pooled Placebo (Cohort C1 to C3): Participants without CF who received placebo matched to VX-445/TEZ/IVA triple combination (TC) once daily in the morning and placebo matched to IVA in the evening for 14 days.
- Part D: Placebo: Participants with CF, F/MF genotype who received placebo matched to VX-445/TEZ/IVA TC once daily in the morning and placebo matched to IVA in the evening for 4 weeks in the TC treatment period.
- Part D: VX-445/TEZ/IVA TC - Low Dose: Participants with CF, F/MF genotype who received VX-445 50 mg qd /TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the TC treatment period.
- Part D: VX-445/TEZ/IVA TC - Medium Dose: Participants with CF, F/MF genotype who received VX-445 100 mg qd /TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the TC treatment period.
- Part D: VX-445/TEZ/IVA TC - High Dose: Participants with CF, F/MF genotype who received VX-445 200 mg qd /TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the TC treatment period.
Period: Overall Study
Arm/Group | Part A: Pooled Placebo (Except Cohort A7) | Part A: VX-445 (Except Cohort A7) | Part A: VX-445 (Cohort A7) | Part B: Pooled Placebo (Cohort B1 to B4) | Part B: VX-445 (Cohort B1 to B4) | Part C: Pooled Placebo (Cohort C1 to C3) | Part C: VX-445/TEZ/IVA TC (Cohort C1 to C3) | Part D: Placebo | Part D: VX-445/TEZ/IVA TC - Low Dose | Part D: VX-445/TEZ/IVA TC - Medium Dose | Part D: VX-445/TEZ/IVA TC - High Dose | Part E: TEZ/IVA | Part E: VX-445/TEZ/IVA TC | Part F: Placebo | Part F: VX-445/TEZ/VX-561 TC
Started | 9 | 30 | 8 | 7 | 25 | 6 | 17 | 12 | 10 | 22 | 21 | 7 | 21 | 8 | 22
Safety Set (Received at least 1 dose of study drug.) | 9 | 30 | 8 | 7 | 25 | 6 | 17 | 12 | 10 | 22 | 21 | 7 | 21 | 8 | 21
Completed | 9 | 30 | 8 | 7 | 24 | 6 | 17 | 12 | 10 | 22 | 21 | 7 | 20 | 8 | 21
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Randomized, Never Dosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part A: VX-445 (Except Cohort A7): Participants without CF who received single ascending dose of VX-445 tablet starting from 20 mg to 360 mg in Cohort A1 to A5.
- Part A: VX-445 (Cohort A7): Participants without CF who received single dose of VX-445 100 mg tablet on Day 1 in fasted state and on Day 7 in fed state, followed by VX-445 20 mg IV injection on Day 13 in fed state in Cohort A7.
- Part B: Pooled Placebo (Cohort B1 to B4): Participants without CF who received multiple doses of placebo matched to VX-445 qd for 10 days in Cohort B1 to B4.
- Part C: Pooled Placebo (Cohort C1 to C3): Participants without CF who received placebo matched to VX-445/TEZ/IVA TC qd in the morning and placebo matched to IVA in the evening for 14 days.
- Part D: Placebo: Participants with CF, F/MF genotype who received placebo matched to VX-445/TEZ/IVA TC qd in the morning and placebo matched to IVA in the evening for 4 weeks in the TC treatment period.
- Part E: VX-445/TEZ/IVA TC: Following run-in period of 4 weeks with TEZ/IVA, participants with CF, F/F genotype who received VX-445 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks in the TC treatment period.
- Total: Total of all reporting groups
Arm/Group | Part A: Pooled Placebo (Except Cohort A7) | Part A: VX-445 (Except Cohort A7) | Part A: VX-445 (Cohort A7) | Part B: Pooled Placebo (Cohort B1 to B4) | Part B: VX-445 (Cohort B1 to B4) | Part C: Pooled Placebo (Cohort C1 to C3) | Part C: VX-445/TEZ/IVA TC (Cohort C1 to C3) | Part D: Placebo | Part D: VX-445/TEZ/IVA TC - Low Dose | Part D: VX-445/TEZ/IVA TC - Medium Dose | Part D: VX-445/TEZ/IVA TC - High Dose | Part E: TEZ/IVA | Part E: VX-445/TEZ/IVA TC | Part F: Placebo | Part F: VX-445/TEZ/VX-561 TC | Total
Number analyzed (Participants) | 9 | 30 | 8 | 7 | 25 | 6 | 17 | 12 | 10 | 22 | 21 | 7 | 21 | 8 | 21 | 224
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 30 | 8 | 7 | 25 | 6 | 17 | 12 | 10 | 22 | 21 | 7 | 21 | 8 | 21 | 224
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 0 | 3 | 0 | 0 | 2 | 6 | 7 | 11 | 1 | 9 | 5 | 10 | 58
  Male | 7 | 28 | 8 | 7 | 22 | 6 | 17 | 10 | 4 | 15 | 10 | 6 | 12 | 3 | 11 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 0 | 1 | 1 | 5 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 13
  Not Hispanic or Latino | 9 | 28 | 6 | 7 | 24 | 5 | 12 | 12 | 10 | 22 | 20 | 7 | 20 | 8 | 20 | 210
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 16 | 4 | 3 | 9 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 42
  White | 5 | 14 | 4 | 2 | 16 | 2 | 16 | 12 | 8 | 22 | 21 | 7 | 21 | 8 | 20 | 178
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Parts A, B and C: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From first dose of study drug in treatment period up to safety follow-up (up to 28 days)
Population: Safety Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Pooled Placebo (Except Cohort A7) | Part A: VX-445 (Except Cohort A7) | Part A: VX-445 (Cohort A7) | Part B: Pooled Placebo (Cohort B1 to B4) | Part B: VX-445 (Cohort B1 to B4) | Part C: Pooled Placebo (Cohort C1 to C3) | Part C: VX-445/TEZ/IVA TC (Cohort C1 to C3)
Number analyzed (Participants) | 9 | 30 | 8 | 7 | 25 | 6 | 17
Participants
  Participants with AEs | 0 | 3 | 1 | 2 | 2 | 2 | 5
  Participants with SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Parts D, E and F: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From first dose of study drug in TC treatment period up to 28 days after last dose of study drug (up to 5 weeks)
Population: The Safety Set will include all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part D: VX-445/TEZ/IVA TC: Participants with CF, F/MF genotype who received VX-445/TEZ/IVA TC for 4 weeks in the TC treatment period.
Arm/Group | Part D: Placebo | Part D: VX-445/TEZ/IVA TC | Part E: TEZ/IVA | Part E: VX-445/TEZ/IVA TC | Part F: Placebo | Part F: VX-445/TEZ/VX-561 TC
Number analyzed (Participants) | 12 | 53 | 7 | 21 | 8 | 21
Participants
  Participants with AEs | 12 | 49 | 5 | 19 | 7 | 19
  Participants with SAEs | 2 | 3 | 1 | 0 | 1 | 0

3. Primary Outcome: Part D: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline through Day 29
Population: The full analysis set (FAS) included all randomized participants who carry the intended CFTR allele mutation and have received at least 1 dose of study drug in the TC treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Arm/Group | Part D: Placebo | Part D: VX-445/TEZ/IVA TC - Low Dose | Part D: VX-445/TEZ/IVA TC - Medium Dose | Part D: VX-445/TEZ/IVA TC - High Dose
Number analyzed (Participants) | 12 | 10 | 22 | 21
percentage points | 0.0 (2.0) | 11.1 (2.1) | 7.9 (1.4) | 13.8 (1.4)
Statistical Analysis 1: Comparison: Part D: Placebo; Test type: Other; p = 0.9943, Mixed-effects model for repeated measure — P value within treatment
Statistical Analysis 2: Comparison: Part D: VX-445/TEZ/IVA TC - Low Dose; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure — P value within treatment
Statistical Analysis 3: Comparison: Part D: VX-445/TEZ/IVA TC - Medium Dose; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure — P value within treatment
Statistical Analysis 4: Comparison: Part D: VX-445/TEZ/IVA TC - High Dose; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure — P value within treatment

4. Primary Outcome: Part E: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline through Day 29
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Arm/Group | Part E: TEZ/IVA | Part E: VX-445/TEZ/IVA TC
Number analyzed (Participants) | 7 | 21
percentage points | 0.4 (2.8) | 11.0 (1.5)
Statistical Analysis 1: Comparison: Part E: TEZ/IVA; Test type: Other; p = 0.8869, Mixed-effects model for repeated measure — P value within treatment
Statistical Analysis 2: Comparison: Part E: VX-445/TEZ/IVA TC; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure — P value within treatment

5. Primary Outcome: Part F: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline through Day 29
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Groups:
- Part F: VX-445/TEZ/VX-561 TC: Participants with CF, F/MF genotype who received VX-445 200 mg/TEZ 100 mg/VX-561 150 mg qd for 4 weeks in the TC treatment period.
Arm/Group | Part F: Placebo | Part F: VX-445/TEZ/VX-561 TC
Number analyzed (Participants) | 8 | 21
percentage points | 1.2 (2.6) | 11.7 (1.6)
Statistical Analysis 1: Comparison: Part F: Placebo; Test type: Other; p = 0.6407, Mixed-effects model for repeated measure — P value within treatment
Statistical Analysis 2: Comparison: Part F: VX-445/TEZ/VX-561 TC; Test type: Other; p < 0.0001, mixed-effects model for repeated measure — P value within treatment

6. Secondary Outcome: Part A: Maximum Observed Concentration (Cmax) of VX-445
Time Frame: Cohort A1-A5: Pre-dose to 96 hours post-dose; Cohort A7: Pre-dose to 120 hours post-dose
Population: The Pharmacokinetic Set included all participants who received at least 1 dose of study drug and for whom the primary PK data are considered sufficient and interpretable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter
Groups:
- Part A: VX-445 (Cohort A1): Participants received single dose of VX-445 20 mg tablet in Cohort A1.
- Part A: VX-445 (Cohort A2): Participants received single dose of VX-445 60 mg tablet in Cohort A2.
- Part A: VX-445 (Cohort A3): Participants received single dose of VX-445 120 mg tablet in Cohort A3.
- Part A: VX-445 (Cohort A4): Participants received single dose of VX-445 240 mg tablet in Cohort A4.
- Part A: VX-445 (Cohort A5): Participants received single dose of VX-445 360 mg tablet in Cohort A5.
- Part A: VX-445 (Cohort A7-Fasted): Participants received single dose of VX-445 100 mg tablet on Day 1 in fasted state in Cohort A7.
- Part A: VX-445 (Cohort A7-Fed): Participants received single dose of VX-445 100 mg tablet on Day 7 in fed state in Cohort A7.
- Part A: VX-445 (Cohort A7-IV): Participants received single IV injection of VX-445 20 mg on Day 13 in fed state in Cohort A7.
Arm/Group | Part A: VX-445 (Cohort A1) | Part A: VX-445 (Cohort A2) | Part A: VX-445 (Cohort A3) | Part A: VX-445 (Cohort A4) | Part A: VX-445 (Cohort A5) | Part A: VX-445 (Cohort A7-Fasted) | Part A: VX-445 (Cohort A7-Fed) | Part A: VX-445 (Cohort A7-IV)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 7 | 7
microgram per milliliter | 0.398 (23.0) | 0.989 (35.1) | 2.52 (13.0) | 4.56 (28.2) | 7.07 (19.1) | 0.486 (27.4) | 1.76 (14.6) | 0.740 (27.1)

7. Secondary Outcome: Part A: Area Under Plasma Concentration Time Curve From Time of Dosing to Last Measurable Concentration (AUC0-tlast) of VX-445
Time Frame: Cohort A1-5: Pre-dose to 96 hours post-dose; Cohort A7: Pre-dose to 120 hours post-dose
Population: The Pharmacokinetic Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter
Arm/Group | Part A: VX-445 (Cohort A1) | Part A: VX-445 (Cohort A2) | Part A: VX-445 (Cohort A3) | Part A: VX-445 (Cohort A4) | Part A: VX-445 (Cohort A5) | Part A: VX-445 (Cohort A7-Fasted) | Part A: VX-445 (Cohort A7-Fed) | Part A: VX-445 (Cohort A7-IV)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 7 | 7
microgram*hour per milliliter | 11.4 (34.2) | 30.8 (21.2) | 87.1 (39.9) | 125 (34.2) | 286 (9.30) | 21.8 (31.5) | 55.1 (14.9) | 13.6 (19.7)

8. Secondary Outcome: Part B: Maximum Observed Concentration (Cmax) of VX-445
Time Frame: Pre-dose to 96 hours post-dose on Day 1 and Day 10
Population: The Pharmacokinetic Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter
Groups:
- Part B: VX-445 (Cohort B1): Participants received VX-445 60 mg tablet once daily for 10 days in Cohort B1.
- Part B: VX-445 (Cohort B2): Participants received VX-445 120 mg tablet once daily for 10 days in Cohort B2.
- Part B: VX-445 (Cohort B3): Participants received VX-445 240 mg tablet once daily for 10 days in Cohort B3.
- Part B: VX-445 (Cohort B4): Participants received VX-445 340 mg tablet once daily for 10 days in Cohort B4.
Arm/Group | Part B: VX-445 (Cohort B1) | Part B: VX-445 (Cohort B2) | Part B: VX-445 (Cohort B3) | Part B: VX-445 (Cohort B4)
Number analyzed (Participants) | 6 | 6 | 6 | 6
microgram per milliliter
  Day 1 | 1.18 (19.9) | 2.82 (25.5) | 3.47 (52.9) | 9.56 (65.6)
  Day 10 | 2.13 (15) | 5.83 (28.1) | 11.4 (27.2) | 18.2 (29.5)

9. Secondary Outcome: Part B: Area Under Plasma Concentration Time Curve From Time of Dosing to Last Measurable Concentration (AUC0-tlast) of VX-445
Time Frame: Pre-dose to 96 hours post-dose on Day 1 and Day 10
Population: The Pharmacokinetic Set. Here "Number analyzed" signifies those participants who were evaluated for this outcome measure at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter
Arm/Group | Part B: VX-445 (Cohort B1) | Part B: VX-445 (Cohort B2) | Part B: VX-445 (Cohort B3) | Part B: VX-445 (Cohort B4)
Number analyzed (Participants) | 6 | 6 | 6 | 6
microgram*hour per milliliter
  Day 1 | 17.9 (20.0) | 42.2 (19.5) | 57.9 (42.8) | 119 (27.5)
  Day 10: number analyzed (Participants) | 6 | 6 | 5 | 6
  Day 10 | 61.4 (21.8) | 183 (32.7) | 452 (41.5) | 692 (47.6)

10. Secondary Outcome: Part B: Observed Pre-dose Plasma Concentration (Ctrough) of VX-445
Time Frame: Pre-dose on Day 10
Population: The Pharmacokinetic Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter
Arm/Group | Part B: VX-445 (Cohort B1) | Part B: VX-445 (Cohort B2) | Part B: VX-445 (Cohort B3) | Part B: VX-445 (Cohort B4)
Number analyzed (Participants) | 6 | 6 | 6 | 6
microgram per milliliter | 1.05 (24.5) | 2.81 (33.2) | 7.10 (30.1) | 11.5 (32.0)

11. Secondary Outcome: Part C: Maximum Observed Concentration (Cmax) of VX-445, TEZ and Its Metabolites (M1-TEZ and M2-TEZ)
Time Frame: Pre-dose to 96 hours post-dose on Day 1, Day 7 and Day 14
Population: The Pharmacokinetic Set. Here "Number analyzed" signified those subjects who were evaluated at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter
Groups:
- Part C: VX-445/TEZ/IVA TC (Cohort C1): Participants received VX-445 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in cohort C1 for 14 days.
- Part C: VX-445/TEZ/IVA TC (Cohort C2): Participants received VX-445 280 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in cohort C2 for 14 days.
- Part C: VX-445/TEZ/IVA TC (Cohort C3): Participants received VX-445 100 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in cohort C3 for 14 days.
Arm/Group | Part C: VX-445/TEZ/IVA TC (Cohort C1) | Part C: VX-445/TEZ/IVA TC (Cohort C2) | Part C: VX-445/TEZ/IVA TC (Cohort C3)
Number analyzed (Participants) | 5 | 6 | 6
microgram per milliliter
  VX-445: Day 1 | 3.04 (23.2) | 4.86 (25.4) | 1.72 (16.5)
  VX-445: Day 7 | 8.29 (31.9) | 10.3 (18.4) | 3.58 (14.8)
  VX-445: Day 14: number analyzed (Participants) | 4 | 6 | 6
  VX-445: Day 14 | 8.71 (9.65) | 14.0 (19.2) | 4.73 (15.9)
  TEZ: Day 1 | 3.81 (16.4) | 5.67 (17.2) | 5.38 (19.2)
  TEZ: Day 7 | 7.09 (19.4) | 8.29 (13.6) | 7.01 (14.7)
  TEZ: Day 14: number analyzed (Participants) | 4 | 6 | 6
  TEZ: Day 14 | 8.11 (21.2) | 9.07 (7.60) | 8.60 (12.8)
  M1-TEZ: Day 1 | 0.929 (35) | 0.988 (31.7) | 1.30 (17.3)
  M1-TEZ: Day 7 | 4.34 (28.7) | 5.19 (16.8) | 5.86 (11.3)
  M1-TEZ: Day 14: number analyzed (Participants) | 4 | 6 | 6
  M1-TEZ: Day 14 | 5.77 (24.6) | 6.79 (14.9) | 7.54 (11.8)
  M2-TEZ: Day 1 | 0.553 (47.0) | 0.667 (39.6) | 0.716 (17.0)
  M2-TEZ: Day 7 | 4.72 (30.3) | 6.41 (33.2) | 5.46 (29.4)
  M2-TEZ: Day 14: number analyzed (Participants) | 4 | 6 | 6
  M2-TEZ: Day 14 | 7.69 (23.7) | 10.1 (24.2) | 7.93 (28.3)

12. Secondary Outcome: Part C: Area Under Plasma Concentration Time Curve From Time of Dosing to Last Measurable Concentration (AUC0-tlast) of VX-445, TEZ and Its Metabolites (M1-TEZ and M2-TEZ)
Time Frame: Pre-dose to 96 hours post-dose on Day 1, Day 7 and Day 14
Population: The Pharmacokinetic Set. Here "Number analyzed" signified those subjects who were evaluated at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter
Arm/Group | Part C: VX-445/TEZ/IVA TC (Cohort C1) | Part C: VX-445/TEZ/IVA TC (Cohort C2) | Part C: VX-445/TEZ/IVA TC (Cohort C3)
Number analyzed (Participants) | 5 | 6 | 6
microgram*hour per milliliter
  VX-445: Day 1 | 48.6 (22.7) | 72.5 (20.7) | 26.4 (13.8)
  VX-445: Day 7 | 156 (37.1) | 177 (30.0) | 65.4 (20.7)
  VX-445: Day 14: number analyzed (Participants) | 4 | 6 | 6
  VX-445: Day 14 | 345 (30.7) | 506 (31.5) | 183 (18.8)
  TEZ: Day 1 | 41.4 (27.5) | 43.8 (9.91) | 42.7 (20.9)
  TEZ: Day 7 | 103 (35.8) | 105 (16.5) | 96.9 (18.9)
  TEZ: Day 14: number analyzed (Participants) | 4 | 6 | 6
  TEZ: Day 14 | 252 (35.1) | 288 (13.6) | 275 (19.5)
  M1-TEZ: Day 1 | 17.7 (37.2) | 20.1 (35.2) | 25.5 (19.1)
  M1-TEZ: Day 7 | 90.9 (29.9) | 110 (17.8) | 125 (14.1)
  M1-TEZ: Day 14: number analyzed (Participants) | 4 | 6 | 6
  M1-TEZ: Day 14 | 380 (22.1) | 477 (16.0) | 512 (17.9)
  M2-TEZ: Day 1 | 6.65 (48.6) | 8.19 (52.5) | 9.00 (16.6)
  M2-TEZ: Day 7 | 108 (31.2) | 143 (34.1) | 123 (28.7)
  M2-TEZ: Day 14: number analyzed (Participants) | 4 | 6 | 6
  M2-TEZ: Day 14 | 617 (23.2) | 831 (29.5) | 652 (31.2)

13. Secondary Outcome: Part C: Maximum Observed Concentration (Cmax) of IVA and Its Metabolites (M1-IVA and M6-IVA)
Time Frame: Pre-dose to 96 hours post-dose on Day 1, Day 7 and Day 14
Population: The Pharmacokinetic Set. Here "Number analyzed" signified those subjects who were evaluated at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Part C: VX-445/TEZ/IVA TC (Cohort C1) | Part C: VX-445/TEZ/IVA TC (Cohort C2) | Part C: VX-445/TEZ/IVA TC (Cohort C3)
Number analyzed (Participants) | 5 | 6 | 6
nanogram per milliliter
  IVA: Day 1 | 425 (29.8) | 461 (49.3) | 437 (9.63)
  IVA: Day 7 | 1290 (41.1) | 1190 (42.4) | 1070 (20.0)
  IVA: Day 14: number analyzed (Participants) | 4 | 6 | 6
  IVA: Day 14 | 1360 (21.9) | 1920 (33.7) | 1410 (25.5)
  M1-IVA: Day 1 | 1250 (29.9) | 1190 (28.1) | 1070 (28.6)
  M1-IVA: Day 7 | 2460 (26.8) | 2590 (28.1) | 2070 (23.1)
  M1-IVA: Day 14: number analyzed (Participants) | 4 | 6 | 6
  M1-IVA: Day 14 | 2680 (19.4) | 3900 (21.4) | 2990 (28.3)
  M6-IVA: Day 1 | 901 (38.2) | 1180 (16.6) | 631 (31.1)
  M6-IVA: Day 7 | 1960 (38.1) | 2590 (7.3) | 1400 (29.8)
  M6-IVA: Day 14: number analyzed (Participants) | 4 | 6 | 6
  M6-IVA: Day 14 | 2060 (30.1) | 3350 (17.4) | 1980 (34.7)

14. Secondary Outcome: Part C: Area Under Plasma Concentration Time Curve From Time of Dosing to Last Measurable Concentration (AUC0-tlast) of IVA and Its Metabolites (M1-IVA and M6-IVA)
Time Frame: Pre-dose to 96 hours post-dose on Day 1, Day 7 and Day 14
Population: The Pharmacokinetic Set. Here "Number analyzed" signified those subjects who were evaluated at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Part C: VX-445/TEZ/IVA TC (Cohort C1) | Part C: VX-445/TEZ/IVA TC (Cohort C2) | Part C: VX-445/TEZ/IVA TC (Cohort C3)
Number analyzed (Participants) | 5 | 6 | 6
nanogram*hour per milliliter
  IVA: Day 1 | 6350 (40.9) | 6210 (45.5) | 5480 (28.5)
  IVA: Day 7 | 21600 (65.6) | 18800 (50.7) | 16900 (28.4)
  IVA: Day 14: number analyzed (Participants) | 4 | 6 | 6
  IVA: Day 14 | 27900 (48.7) | 35000 (44.8) | 32600 (40.6)
  M1-IVA: Day 1 | 16900 (38.9) | 14800 (32.3) | 13300 (21.1)
  M1-IVA: Day 7 | 47500 (43.6) | 46300 (30.6) | 36400 (25.9)
  M1-IVA: Day 14: number analyzed (Participants) | 4 | 6 | 6
  M1-IVA: Day 14 | 75300 (42.7) | 97000 (31.3) | 86100 (30.2)
  M6-IVA: Day 1 | 11100 (49.9) | 14100 (20.3) | 9050 (26.1)
  M6-IVA: Day 7 | 39700 (38.8) | 51400 (13.0) | 29100 (36.0)
  M6-IVA: Day 14: number analyzed (Participants) | 4 | 6 | 6
  M6-IVA: Day 14 | 66300 (44.9) | 123000 (23.1) | 67100 (42.3)

15. Secondary Outcome: Part C: Observed Pre-dose Concentration (Ctrough) of VX-445, TEZ and Its Metabolites (M1-TEZ and M2-TEZ)
Time Frame: Pre-dose on Day 7 and Day 14
Population: The Pharmacokinetic Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter
Arm/Group | Part C: VX-445/TEZ/IVA TC (Cohort C1) | Part C: VX-445/TEZ/IVA TC (Cohort C2) | Part C: VX-445/TEZ/IVA TC (Cohort C3)
Number analyzed (Participants) | 5 | 6 | 6
microgram per milliliter
  VX-445: Day 7 | 4.63 (46.8) | 5.91 (35.5) | 2.09 (14.9)
  VX-445: Day 14 | 4.45 (38.9) | 7.60 (29.8) | 2.92 (13.2)
  TEZ: Day 7 | 2.73 (48.7) | 2.77 (19.2) | 2.52 (23.0)
  TEZ: Day 14 | 3.10 (33.4) | 3.70 (16.0) | 3.62 (24.6)
  M1-TEZ: Day 7 | 3.36 (27.1) | 3.98 (16.8) | 4.71 (14.0)
  M1-TEZ: Day 14 | 4.38 (20.5) | 5.42 (16.1) | 5.52 (12.9)
  M2-TEZ: Day 7 | 4.06 (32.8) | 5.63 (37.5) | 4.92 (27.7)
  M2-TEZ: Day 14 | 6.46 (22.5) | 8.85 (29.9) | 7.38 (29.6)

16. Secondary Outcome: Part C: Observed Pre-dose Concentration (Ctrough) of IVA and Its Metabolites (M1-IVA and M6-IVA)
Time Frame: Pre-dose on Day 7 and Day 14
Population: The Pharmacokinetic Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Part C: VX-445/TEZ/IVA TC (Cohort C1) | Part C: VX-445/TEZ/IVA TC (Cohort C2) | Part C: VX-445/TEZ/IVA TC (Cohort C3)
Number analyzed (Participants) | 5 | 6 | 6
nanogram per milliliter
  IVA: Day 7 | 753 (75) | 759 (45.7) | 604 (32.8)
  IVA: Day 14 | 610 (55.6) | 990 (43.4) | 881 (35.3)
  M1-IVA: Day 7 | 1790 (43.7) | 1960 (21.4) | 1400 (21.3)
  M1-IVA: Day 14 | 1600 (46.2) | 2210 (19.8) | 1930 (16.9)
  M6-IVA: Day 7 | 1530 (31.5) | 2260 (11.9) | 1270 (32.1)
  M6-IVA: Day 14 | 1360 (49.1) | 2600 (18.0) | 1640 (27.0)

17. Secondary Outcome: Part D: Observed Pre-dose Plasma Concentration (Ctrough) of VX-445, TEZ and Its Metabolite (M1-TEZ), IVA and Its Metabolite (M1-IVA)
Time Frame: Pre-dose on Day 15 and Day 29
Population: FAS. Here "number analyzed" signifies those participants who were evaluated at specified time points for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Part D: VX-445/TEZ/IVA TC - Low Dose | Part D: VX-445/TEZ/IVA TC - Medium Dose | Part D: VX-445/TEZ/IVA TC - High Dose
Number analyzed (Participants) | 10 | 21 | 21
microgram per milliliter
  VX-445: Day 15: number analyzed (Participants) | 10 | 21 | 20
  VX-445: Day 15 | 1.04 (0.612) | 2.15 (0.977) | 5.77 (4.14)
  VX-445: Day 29 | 1.27 (0.530) | 2.18 (1.26) | 5.57 (2.80)
  TEZ: Day 15: number analyzed (Participants) | 10 | 21 | 20
  TEZ: Day 15 | 1.85 (1.26) | 1.68 (0.700) | 1.76 (0.960)
  TEZ: Day 29 | 2.16 (1.27) | 1.77 (0.833) | 2.22 (1.62)
  M1-TEZ: Day 15: number analyzed (Participants) | 10 | 21 | 20
  M1-TEZ: Day 15 | 4.46 (1.96) | 4.11 (1.47) | 4.43 (1.79)
  M1-TEZ: Day 29 | 4.77 (2.04) | 4.30 (1.55) | 4.74 (1.89)
  IVA: Day 15: number analyzed (Participants) | 10 | 21 | 20
  IVA: Day 15 | 0.720 (0.484) | 0.665 (0.414) | 0.701 (0.593)
  IVA: Day 29 | 0.753 (0.424) | 0.704 (0.414) | 0.658 (0.386)
  M1-IVA: Day 15: number analyzed (Participants) | 10 | 21 | 20
  M1-IVA: Day 15 | 1.29 (0.748) | 1.21 (0.666) | 1.45 (1.22)
  M1-IVA: Day 29: number analyzed (Participants) | 10 | 20 | 21
  M1-IVA: Day 29 | 1.57 (0.830) | 1.20 (0.717) | 1.29 (0.797)

18. Secondary Outcome: Part E: Observed Pre-dose Concentration (Ctrough) of VX-445, TEZ and Its Metabolite (M1-TEZ) and IVA and Its Metabolite (M1-IVA)
Time Frame: Pre-dose on Day 15 and Day 29
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Part E: TEZ/IVA | Part E: VX-445/TEZ/IVA TC
Number analyzed (Participants) | 7 | 21
microgram per milliliter
  VX-445: Day 15: number analyzed (Participants) | 0 | 21
  VX-445: Day 15 |  | 5.07 (2.47)
  VX-445: Day 29: number analyzed (Participants) | 0 | 20
  VX-445: Day 29 |  | 5.35 (3.73)
  TEZ: Day 15 | 1.85 (0.863) | 1.86 (1.09)
  TEZ: Day 29: number analyzed (Participants) | 7 | 20
  TEZ: Day 29 | 1.84 (1.28) | 1.99 (1.55)
  M1-TEZ: Day 15 | 3.96 (1.76) | 4.57 (1.73)
  M1-TEZ: Day 29: number analyzed (Participants) | 7 | 20
  M1-TEZ: Day 29 | 3.73 (1.51) | 4.71 (1.86)
  IVA: Day 15 | 0.766 (0.366) | 0.659 (0.529)
  IVA: Day 29: number analyzed (Participants) | 7 | 20
  IVA: Day 29 | 0.595 (0.303) | 0.798 (0.901)
  M1-IVA: Day 15 | 1.22 (0.470) | 1.09 (0.973)
  M1-IVA: Day 29: number analyzed (Participants) | 7 | 20
  M1-IVA: Day 29 | 0.943 (0.431) | 1.43 (1.54)

19. Secondary Outcome: Part F: Observed Pre-dose Concentration (Ctrough) of VX-445, TEZ and Its Metabolite (M1-TEZ) and VX-561
Time Frame: Pre-dose on Day 15 and Day 29
Population: FAS. Here, "Number analyzed" signifies those participants who were evaluated at specified time points for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Part F: VX-445/TEZ/VX-561 TC
Number analyzed (Participants) | 20
microgram per milliliter
  VX-445: Day 15: number analyzed (Participants) | 19
  VX-445: Day 15 | 4.40 (1.54)
  VX-445: Day 29 | 5.25 (2.88)
  TEZ: Day 15: number analyzed (Participants) | 19
  TEZ: Day 15 | 1.80 (0.658)
  TEZ: Day 29 | 2.22 (1.65)
  M1-TEZ: Day 15: number analyzed (Participants) | 19
  M1-TEZ: Day 15 | 4.99 (1.71)
  M1-TEZ: Day 29 | 5.09 (1.37)
  VX-561: Day 15: number analyzed (Participants) | 19
  VX-561: Day 15 | 0.441 (0.174)
  VX-561: Day 29 | 0.597 (0.473)

20. Secondary Outcome: Part D: Absolute Change in Sweat Chloride Concentration
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline through Day 29
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Part D: Placebo | Part D: VX-445/TEZ/IVA TC - Low Dose | Part D: VX-445/TEZ/IVA TC - Medium Dose | Part D: VX-445/TEZ/IVA TC - High Dose
Number analyzed (Participants) | 12 | 10 | 22 | 21
millimole per liter (mmol/L) | -2.2 (3.9) | -38.2 (4.2) | -33.2 (2.8) | -39.1 (2.9)
Statistical Analysis 1: Comparison: Part D: Placebo; Test type: Other; p = 0.5802, Mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 2: Comparison: Part D: VX-445/TEZ/IVA TC - Low Dose; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 3: Comparison: Part D: VX-445/TEZ/IVA TC - Medium Dose; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 4: Comparison: Part D: VX-445/TEZ/IVA TC - High Dose; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control

21. Secondary Outcome: Part E: Absolute Change in Sweat Chloride Concentration
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline through Day 29
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Part E: TEZ/IVA | Part E: VX-445/TEZ/IVA TC
Number analyzed (Participants) | 7 | 21
mmol/L | 0.8 (4.9) | -39.6 (2.8)
Statistical Analysis 1: Comparison: Part E: TEZ/IVA; Test type: Other; p = 0.8712, mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 2: Comparison: Part E: VX-445/TEZ/IVA TC; Test type: Other; p < 0.0001, mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control

22. Secondary Outcome: Part F: Absolute Change in Sweat Chloride Concentration
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline through Day 29
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Part F: Placebo | Part F: VX-445/TEZ/VX-561 TC
Number analyzed (Participants) | 8 | 21
mmol/L | 1.0 (4.6) | -33.6 (2.8)
Statistical Analysis 1: Comparison: Part F: Placebo; Test type: Other; p = 0.8359, mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 2: Comparison: Part F: VX-445/TEZ/VX-561 TC; Test type: Other; p < 0.0001, mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control

23. Secondary Outcome: Part D: Relative Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline through Day 29
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part D: Placebo | Part D: VX-445/TEZ/IVA TC - Low Dose | Part D: VX-445/TEZ/IVA TC - Medium Dose | Part D: VX-445/TEZ/IVA TC - High Dose
Number analyzed (Participants) | 12 | 10 | 22 | 21
percent change | 0.3 (4.0) | 19.3 (4.2) | 13.8 (2.8) | 26.2 (2.9)
Statistical Analysis 1: Comparison: Part D: Placebo; Test type: Other; p = 0.9453, Mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 2: Comparison: Part D: VX-445/TEZ/IVA TC - Low Dose; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 3: Comparison: Part D: VX-445/TEZ/IVA TC - Medium Dose; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 4: Comparison: Part D: VX-445/TEZ/IVA TC - High Dose; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control

24. Secondary Outcome: Part E: Relative Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline through Day 29
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part E: TEZ/IVA | Part E: VX-445/TEZ/IVA TC
Number analyzed (Participants) | 7 | 21
percent change | 1.4 (5.0) | 19.2 (2.7)
Statistical Analysis 1: Comparison: Part E: TEZ/IVA; Test type: Other; p = 0.7849, mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 2: Comparison: Part E: VX-445/TEZ/IVA TC; Test type: Other; p < 0.0001, mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control

25. Secondary Outcome: Part F: Relative Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline through Day 29
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part F: Placebo | Part F: VX-445/TEZ/VX-561 TC
Number analyzed (Participants) | 8 | 21
percent change | 1.6 (4.6) | 19.9 (2.8)
Statistical Analysis 1: Comparison: Part F: Placebo; Test type: Other; p = 0.7356, mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 2: Comparison: Part F: VX-445/TEZ/VX-561 TC; Test type: Other; p < 0.0001, mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control

26. Secondary Outcome: Part D: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline through Day 29
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Part D: Placebo | Part D: VX-445/TEZ/IVA TC - Low Dose | Part D: VX-445/TEZ/IVA TC - Medium Dose | Part D: VX-445/TEZ/IVA TC - High Dose
Number analyzed (Participants) | 12 | 10 | 22 | 21
units on a scale | 4.2 (4.9) | 20.8 (5.4) | 15.4 (3.7) | 25.7 (3.7)
Statistical Analysis 1: Comparison: Part D: Placebo; Test type: Other; p = 0.3940, Mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 2: Comparison: Part D: VX-445/TEZ/IVA TC - Low Dose; Test type: Other; p = 0.0003, Mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 3: Comparison: Part D: VX-445/TEZ/IVA TC - Medium Dose; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 4: Comparison: Part D: VX-445/TEZ/IVA TC - High Dose; Test type: Other; p < 0.0001, Mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control

27. Secondary Outcome: Part E: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: as for outcome 26
Time Frame: From Baseline through Day 29
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Part E: TEZ/IVA | Part E: VX-445/TEZ/IVA TC
Number analyzed (Participants) | 7 | 21
units on a scale | 5.2 (7.1) | 20.7 (4.0)
Statistical Analysis 1: Comparison: Part E: TEZ/IVA; Test type: Other; p = 0.4757, mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 2: Comparison: Part E: VX-445/TEZ/IVA TC; Test type: Other; p < 0.0001, mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control

28. Secondary Outcome: Part F: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: as for outcome 26
Time Frame: From Baseline through Day 29
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Part F: Placebo | Part F: VX-445/TEZ/VX-561 TC
Number analyzed (Participants) | 8 | 21
units on a scale | 20.2 (6.9) | 20.2 (4.3)
Statistical Analysis 1: Comparison: Part F: Placebo; Test type: Other; p = 0.0070, mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control
Statistical Analysis 2: Comparison: Part F: VX-445/TEZ/VX-561 TC; Test type: Other; p < 0.0001, mixed-effects model for repeated measure — P value within treatment. These are nominal p-values without multiplicity control

ADVERSE EVENTS:
Time Frame: Parts A, B and C: From first dose of study drug in treatment period up to safety follow-up (up to 28 days); Parts D, E and F: From first dose of study drug in TC treatment period up to 28 days after last dose of study drug (up to 5 weeks)
Description: MedDRA version 19.1 for Parts A, B and C and MedDRA version 20.1 for Parts D, E and F.
Groups:
- Part C: Pooled Placebo (Cohort C1 to C3): Participants without CF who received placebo matched to VX-445/TEZ/IVA TC once daily in the morning and placebo matched to IVA in the evening for 14 days.
Arm/Group | Part A: Pooled Placebo (Except Cohort A7) | Part A: VX-445 (Except Cohort A7) | Part A: VX-445 (Cohort A7) | Part B: Pooled Placebo (Cohort B1 to B4) | Part B: VX-445 (Cohort B1 to B4) | Part C: Pooled Placebo (Cohort C1 to C3) | Part C: VX-445/TEZ/IVA TC (Cohort C1 to C3) | Part D: Placebo | Part D: VX-445/TEZ/IVA TC - Low Dose | Part D: VX-445/TEZ/IVA TC - Medium Dose | Part D: VX-445/TEZ/IVA TC - High Dose | Part E: TEZ/IVA | Part E: VX-445/TEZ/IVA TC | Part F: Placebo | Part F: VX-445/TEZ/VX-561 TC
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/30 | 0/8 | 0/7 | 0/25 | 0/6 | 0/17 | 0/12 | 0/10 | 0/22 | 0/21 | 0/7 | 0/21 | 0/8 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/30 | 0/8 | 0/7 | 0/25 | 0/6 | 0/17 | 2/12 | 1/10 | 2/22 | 0/21 | 1/7 | 0/21 | 1/8 | 0/21
Other Adverse Events (participants affected / at risk) | 0/9 | 3/30 | 1/8 | 2/7 | 2/25 | 2/6 | 5/17 | 12/12 | 10/10 | 19/22 | 17/21 | 5/7 | 18/21 | 7/8 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Pooled Placebo (Except Cohort A7) (N=9) | Part A: VX-445 (Except Cohort A7) (N=30) | Part A: VX-445 (Cohort A7) (N=8) | Part B: Pooled Placebo (Cohort B1 to B4) (N=7) | Part B: VX-445 (Cohort B1 to B4) (N=25) | Part C: Pooled Placebo (Cohort C1 to C3) (N=6) | Part C: VX-445/TEZ/IVA TC (Cohort C1 to C3) (N=17) | Part D: Placebo (N=12) | Part D: VX-445/TEZ/IVA TC - Low Dose (N=10) | Part D: VX-445/TEZ/IVA TC - Medium Dose (N=22) | Part D: VX-445/TEZ/IVA TC - High Dose (N=21) | Part E: TEZ/IVA (N=7) | Part E: VX-445/TEZ/IVA TC (N=21) | Part F: Placebo (N=8) | Part F: VX-445/TEZ/VX-561 TC (N=21)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza A virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jugular vein thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Pooled Placebo (Except Cohort A7) (N=9) | Part A: VX-445 (Except Cohort A7) (N=30) | Part A: VX-445 (Cohort A7) (N=8) | Part B: Pooled Placebo (Cohort B1 to B4) (N=7) | Part B: VX-445 (Cohort B1 to B4) (N=25) | Part C: Pooled Placebo (Cohort C1 to C3) (N=6) | Part C: VX-445/TEZ/IVA TC (Cohort C1 to C3) (N=17) | Part D: Placebo (N=12) | Part D: VX-445/TEZ/IVA TC - Low Dose (N=10) | Part D: VX-445/TEZ/IVA TC - Medium Dose (N=22) | Part D: VX-445/TEZ/IVA TC - High Dose (N=21) | Part E: TEZ/IVA (N=7) | Part E: VX-445/TEZ/IVA TC (N=21) | Part F: Placebo (N=8) | Part F: VX-445/TEZ/VX-561 TC (N=21)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 3 | 1 | 1 | 1 | 3 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 4 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 2 | 2 | 2 | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 5 | 7 | 1 | 7 | 2 | 5
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 4 | 5 | 0 | 8 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 2 | 0 | 3 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 1 | 1 | 3 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary function test decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 4 | 2 | 0 | 5 | 3 | 3
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT03227471/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT03227471/SAP_001.pdf